CLINICAL TRIAL: NCT02801513
Title: Maintaining Mechanisms of Chronic Depression and Their Changeability: the Role of Discrepancy-based Processing
Brief Title: Maintaining Mechanisms of Chronic Depression and Their Changeability
Acronym: GetWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Freie Universität Berlin (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Thorsten Barnhofer, Heisenberg-Fellow, Freie Universität Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BA2255/3-1
Record Dates: First submitted 2016-06-11; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Major Depressive Disorder
Keywords: mindfulness; EEG; error-related negativity; late positive potential; long-range temporal correlations
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Mindfulness Training (Experimental): The brief mindfulness training comprised of three 1.5-hour weekly individual sessions and included intensive daily home practice. Participants were asked to engage in formal meditation practice for about 25 minutes twice per day on six out of seven days of each week using recorded guided meditations. Practices were shorter in duration than the practices in Mindfulness-Based Cognitive Therapy (MBCT, Segal et al., 2002) in order to allow for more flexibility in scheduling the practices, but followed the standard sequence of mindfulness-based interventions.
  Interventions: Behavioral: Brief Mindfulness Training
- Resting Control Training (Active Comparator): The resting control training comprised of three 1.5-hour weekly individual sessions and included intensive daily home practice. Participants were asked to schedule regular rest periods as a means of deliberately retreating from the activities of the day. Length and frequency of the rest periods mirrored the time demands of the meditation training. Participants received a plausible rationale for the control training that linked acute depression to stress and suggested rest, relaxation, and disengagement from negative thinking as an initial and preliminary step towards recovery.
  Interventions: Behavioral: Resting Control Training

INTERVENTIONS:
Behavioral: Brief Mindfulness Training — Brief mindfulness training comprising of three weekly individual sessions and daily guided meditation home practice
  Other Names: Mindfulness Intervention
  Arms: Brief Mindfulness Training
Behavioral: Resting Control Training — Brief resting control training comprising of three weekly individual sessions and daily home practice consisting of resting periods
  Other Names: Resting Control
  Arms: Resting Control Training

SUMMARY:
Despite considerable progress in the understanding of depression, the treatment of those who have entered a chronic course of the disorder still represents a major challenge. In order to develop more effective interventions it is important to learn more about maintaining mechanisms and the ways in which these can be addressed. Recent research has outlined aberrations in neurophysiological parameters that may serve as risk factors underlying tendencies to engage in maladaptive responses to negative mood, and that may be particularly pronounced in patients with chronic depression. Initial evidence suggests that such deficits may not be easily amenable through established treatments. The current study investigated whether mental training using mindfulness mediation, as compared to an active control training, could alter these parameters in chronically depressed patients.

DETAILED DESCRIPTION:
Persistent engagement in maladaptive patterns of thinking is a hallmark of depression. In those who suffer from a chronic course of the disorders, tendencies towards engagement in such patterns of thinking are likely to have become habitual and automatic in nature. Recent research has begun to elucidate potential cognitive and neurophysiological bases of such persistence. There is evidence that depressed patients show significant deficits in performance monitoring (Weinberg, Dieterich, & Riesel, 2015). Research on error-related negativity (ERN), a signal that occurs briefly after commission of an error, has reported significant aberrations in depressed suggesting deficits at the early stages of processing discrepancies. Deficits in ERN have been suggested to serve as an endophenotype for depression and psychopathology more generally (Manoach & Agam, 2013). Preliminary findings suggest that deficits remain even when symptoms are reduced following established treatments. Similarly, there is evidence for increased tendencies to elaborate negative information as evidenced by stronger late positive potentials (LPP; Auerbach, Stanton, Proudfit, & Pizzagalli, 2015) and an increased rigidity of spontaneous activity of the brain during rest as indicated by increased long-range temporal correlations of spontaneous brain oscillations (LRTC; Bornas et al., 2013).

Interventions using mental training may be particularly suited to address these aberrations. Indeed even brief training in mindfulness has been found to have significant neuroplastic effects (Tang et al., 2010) The aim of the current study was therefore to investigate the effects of a brief intervention using training in mindfulness meditation on the above listed parameters. Chronically depressed patients were randomly allocated to receive either a two-week mindfulness training or a resting control training. EEG was measured before and after the intervention along with self-reports of current symptoms and resilience/vulnerability factors. We expected the mindfulness training to have significantly stronger effects on ERN, LPP, and LRTC than the resting control training.

ELIGIBILITY:
Inclusion Criteria:

* a current diagnosis of Major Depression as assessed by Structured Clinical Interview for DSM IV (First, Spitzer, Gibbon, & Williams, 2002)
* a lifetime history of depression with onset before age 19 and either chronic persistence of symptoms or a history of at least three previous episodes of depression, two of which needed to have occurred during the last two years
* self-reported severity of current symptoms on a clinical level as indicated by Beck Depression Inventory-II (Beck, Steer, & Brown, 1996) scores above 19
* age 25 to 60 thus excluding cases of late-onset depression, and e) fluency in spoken and written German.

Exclusion Criteria:

* history of psychosis or mania, current eating disorder, OCD, current self-harm, current substance abuse or dependence
* history of traumatic brain injury
* current treatment with CBT
* We allowed patients who were currently taking antidepressants into the study provided that the medication had not been changed during the last four weeks before entry into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Error-related negativity | Two weeks
  Event-related potential (EEG)
Long-range temporal correlations of theta oscillations in resting EEG | Two weeks
  Resting EEG
Late positive potentials | Two weeks
  Event-related potential (EEG)

SECONDARY OUTCOMES:
Levels of state mindfulness | Two weeks
  Self-report
Interoceptive awareness | Two weeks
  Self-report
Levels of depressive symptoms | Two weeks
  Self-report
Ruminative tendencies | Two weeks
  Self-report

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Barnhofer, PhD, Principal Investigator — Freie Universität Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auerbach RP, Stanton CH, Proudfit GH, Pizzagalli DA. Self-referential processing in depressed adolescents: A high-density event-related potential study. J Abnorm Psychol. 2015 May;124(2):233-45. doi: 10.1037/abn0000023. Epub 2015 Feb 2. PMID 25643205
- [Background] Bornas, X., Noguera, M., Balle, M., Morillas-Romero, A., Aguayo-Siquier, B., Tortella-Feliu, M., & Llabrés, J. (2013). Long-Range Temporal Correlations in Resting EEG. Journal of Psychophysiology, 27(2), 60-66. doi:10.1027/0269-8803/a000087
- [Background] Manoach DS, Agam Y. Neural markers of errors as endophenotypes in neuropsychiatric disorders. Front Hum Neurosci. 2013 Jul 18;7:350. doi: 10.3389/fnhum.2013.00350. eCollection 2013. PMID 23882201
- [Background] Tang YY, Lu Q, Geng X, Stein EA, Yang Y, Posner MI. Short-term meditation induces white matter changes in the anterior cingulate. Proc Natl Acad Sci U S A. 2010 Aug 31;107(35):15649-52. doi: 10.1073/pnas.1011043107. Epub 2010 Aug 16. PMID 20713717
- [Background] Weinberg A, Dieterich R, Riesel A. Error-related brain activity in the age of RDoC: A review of the literature. Int J Psychophysiol. 2015 Nov;98(2 Pt 2):276-299. doi: 10.1016/j.ijpsycho.2015.02.029. Epub 2015 Mar 4. PMID 25746725
- [Result] Fissler, M. Winnebeck, E., Schroeter, T. A., Gummersbach, M., Huntexburg, J. M., Gaertner, M., & Barnhofer, T. (in press). An Investigation of the Effects of Brief Mindfulness Training on Self-Reported Interoceptive Awareness, the Ability to Decenter, and Their Role in the Reduction of Depressive Symptoms. Mindfulness.
- [Derived] Barnhofer T, Reess TJ, Fissler M, Winnebeck E, Grimm S, Gartner M, Fan Y, Huntenburg JM, Schroeter TA, Gummersbach M, Bajbouj M, Holzel BK. Effects of Mindfulness Training on Emotion Regulation in Patients With Depression: Reduced Dorsolateral Prefrontal Cortex Activation Indexes Early Beneficial Changes. Psychosom Med. 2021 Jul-Aug 01;83(6):579-591. doi: 10.1097/PSY.0000000000000955. PMID 34213860